CLINICAL TRIAL: NCT01101386
Title: Evaluation of Sulfobutylether-ß-cyclodextrin Sodium (SBECD) Accumulation and Voriconazole Pharmacokinetics in Patients Undergoing Continuous Renal Replacement Therapy
Brief Title: Study of Cyclodextrin (SBECD) and Voriconazole Blood Concentrations During Continuous Dialysis
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 10-0136
Record Dates: First submitted 2010-04-06; First posted 2010-04-09 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Fungal Infection
Keywords: Voriconazole; SBECD; pharmacokinetics; Renal Failure
MeSH Terms: conditions — Mycoses; Renal Insufficiency | interventions — Voriconazole

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, urine, effluent fluid from dialysis machine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Voriconazole: Pharmacokinetic Monitoring
  Interventions: Drug: Voriconazole

INTERVENTIONS:
Drug: Voriconazole — Patients will be started on voriconazole 6 mg/kg IV q12h on day 1, then 4 mg/kg IV q12h thereafter.
  Other Names: Vfend

SUMMARY:
This study's primary objective is to determine if continuous renal replacement therapy (CRRT) can adequately remove the sulfobutylether-ß-cyclodextrin sodium (SBECD) vehicle from the blood so that intravenous voriconazole can be utilized in critically ill patients with renal dysfunction requiring dialysis. Secondarily, the pharmacokinetics of intravenous voriconazole and its metabolite (UK121-265) and adverse effects of SBECD accumulation will also be evaluated. The study hypothesis is that CRRT is effective at removing SBECD and allows patients to receive intravenous voriconazole without the concern of SBECD accumulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are receiving continuous renal replacement therapy and are prescribed voriconazole therapy for the treatment or prophylaxis of a fungal infection.

Exclusion Criteria:

* Patients expected to be on CRRT for < 5 days,
* Patients with Child-Pugh C cirrhosis, and
* Patients who are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2010-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Determine SBECD plasma and effluent concentrations | Days 1-7
  Evaluate SBECD pharmacokinetics (Cmax, Cmin, AUC, half-life, CL, seiving coefficient). Predict time to SBECD accumulation in study patients

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Days 1-30
Determine Voriconazole and UK121-265 plasma and effluent concentrations | Days 1-7
  Voriconazole and UK121-265 Pharmacokinetics will be evaluated (Cmax, Cmin, AUC, elimination rate constant, half-life, CL, seiving coefficient) including determination and impact of any CYP2C19 mutations on plasma pharmacokinetic parameters

CONTACTS AND LOCATIONS:
Overall Officials: Ty H Kiser, PharmD, Principal Investigator — Univesity of Colorado Anschutz Medical Campus
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

REFERENCES:
- [Derived] Kiser TH, Fish DN, Aquilante CL, Rower JE, Wempe MF, MacLaren R, Teitelbaum I. Evaluation of sulfobutylether-beta-cyclodextrin (SBECD) accumulation and voriconazole pharmacokinetics in critically ill patients undergoing continuous renal replacement therapy. Crit Care. 2015 Feb 3;19(1):32. doi: 10.1186/s13054-015-0753-8. PMID 25645660